CLINICAL TRIAL: NCT03128086
Title: Protocol-directed Weaning From Mechanical Ventilation in Neurological Patients: a Controlled Trial
Brief Title: Weaning From Mechanical Ventilation in Neurological Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because the principal investigator has moved to another hospital
Sponsor: Hospital General Universitario de Castellón (Other)
Responsible Party: Principal Investigator, ALBERTO BELENGUER MUNCHARAZ, Principal investigator, Hospital General Universitario de Castellón
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HGU Castellon-001
Record Dates: First submitted 2017-03-03; First posted 2017-04-25 (Actual); Results first posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Neurological Diseases or Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protocol-directed weaning (Experimental): A protocol-directed weaning in neurological patients undergoing mechanical ventilation: performing a spontaneous breathing trial through a T-tube and after that to assess the patient's capacity to maintain airway. In case of reach a score the patient will extubated.
  Interventions: Procedure: Protocol-directed weaning
- Conventional weaning (No Intervention): A control group of weaning from mechanical ventilation according to the usual procedure: performing a spontaneous breathing trial through a T-tube and then extubation if the patient success this trial.

INTERVENTIONS:
Procedure: Protocol-directed weaning — A protocol-directed weaning in neurological patients undergoing mechanical ventilation will reduce the rate of extubation failure and associated complications comparing with a conventional weaning (control group)
  Other Names: No other intervention
  Arms: Protocol-directed weaning

SUMMARY:
After a period of mechanical ventilation, a spontaneous breathing trial is performed before extubation in order to assess the patient's ability to breathe. In neurological patients a spontaneous breathing trial can not predict the success of extubation. The extubation failure is associated with a longer intensive care unit stay and hospital stay, as well as more infections and higher mortality.

The purpose of this study is to demonstrate that the use of a protocol-directed weaning in neurological patients reduces the rate of extubation failure and associated complications.

DETAILED DESCRIPTION:
Protocol Patients will be included in the study if they meet the following conditions: no or minimal sedation (Propofol ≤1miligram per kilogram per hour (mg/kg/h) o Midazolam ≤0,1mg/ kg/h), with a spontaneous ventilatory stimulus, absence of intracranial hypertension, Glasgow Coma Score > 9 (with a motor score > 4 points), Noradrenaline ≤ 0,2mcgr/kg/min, fraction of inspired oxygen ≤ 0.5, positive end-expiratory pressure of 5 centimeters of water (cmH20), no scheduled surgery in the next 48 hours, maximal inspiratory pressure < -20 cmH20 (means occlusion pressure test) and a airway occlusion pressure at 0.1 sec (P0.1) >6 millimeters of mercury (mmHg) with a support pressure of 7 cmH20 and 0 cmH20 of positive end-expiratory pressure.

Protocol study (study group). Spontaneous Breathing Trial (SBT). The patient will be connected to mechanical ventilation in a pressure support ventilation mode, which one will be gradually reduced (until a level de pressure support of 10 cmH20 above 5 cmH20 of positive end-expiratory pressure). After, the patient will be disconnected from the ventilator and a spontaneous breathing trial will begin through the connexion of the patient to a T-tube and a source of oxygen. Hemodynamic parameters [systolic blood pressure, heart rate], and breathing parameters [respiratory rate, partial pressure of oxygen, partial pressure of carbonic anhydrid, partial pressure of oxygen to fraction of oxygen ratio, and pH through blood gas analysis and saturation of oxyhemoglobin by pulse oximetry], and neurological (means by Glasgow Coma Score) will be collected during final period of pressure support ventilation (before disconnection) and at onset (5 minutes) and final (between 30 to 120 minutes) of spontaneous breathing trial. A once daily spontaneous breathing trial will be stablished in all the patients until they were extubated. Unsuccessful spontaneous breathing trial will be considered with more than 2 criteria: partial pressure of arterial oxygen of 50-60mmHg with fraction of inspired oxygen ≤ 0.5 (or transcutaneous pulse oximetry <90%), partial pressure of carbonic anhydride > 50 mmHg, pH <7.35, respiratory rate > 35breath per minute, heart rate > 140 beats per minute, systolic blood pressure > 180mmHg, cardiac arrhythmias during spontaneous breathing trial, dyspnea, and increased use of accessory muscles. If the SBT fails, the patient will reconnect to mechanical ventilation. A successful spontaneous breathing trial is defined as absence of whatever of variables above defined.

Airway Patency. Otherwise, if the spontaneous breathing trial is successful, the ability to maintain airway will be analyzed by the following variables: Number of aspirations of secretions/ nursing shift (No aspiration-0, 1 aspiration-1, 2 aspiration-2, ≥ 3 aspiration-3), cough capacity (Strong -0, Mild-1, Weak-2, Absent-3), Appearance and color of secretions: [Viscosity (liquid-0, frothy-1, thick-2, dry-3) and color (clear- 0, brown- 1, yellow-2, green-3)] and the presence of gag reflex (strong- 0, moderate- 1, weak- 2, absent- 3). A score ≤8 is considered as adequate to keep the permeability of airway. Then the patient will be extubated and connected to oxygen mask with fraction of inspired oxygen of 0.4. In case of extubation failure, the patient will be reintubated. The use of non-invasive ventilation is not considered in this study (neither prevention of extubation failure nor in case of extubation failure).

Conventional weaning (control group). Patients in the control group will receive weaning from mechanical ventilation according to the usual procedure, by reducing level of pressure support ventilation. Then a spontaneous breathing trial will be performed through a T-tube (the same parameters as protocol study will collected) and subsequent extubation of the patient if there is a successful spontaneous breathing trial. The criteria for spontaneous breathing trial failure and for extubation failure are the same than in the study group. In case of extubation failure, non-invasive ventilation will be not considered, but it left to the discretion of the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic or hemorrhagic stroke,
* Acute subarachnoid hemorrhage,
* Traumatic brain trauma,
* Metabolic encephalopathy (toxic, infectious as encephalitis or meningitis),
* Scheduled neurosurgical surgery with a prolonged mechanical ventilation
* Status epilepticus
* No or minimal sedation (Propofol ≤1mg/kg/h o Midazolam ≤0,1mg/ kg/h),
* A spontaneous ventilatory stimulus,
* Absence of intracranial hypertension,
* Glasgow Coma Score > 9 (with a motor score > 4 points),
* Noradrenaline ≤ 0,2mcgr/kg/min,
* Fraction of inspired oxygen ≤ 0.5 with a positive end-expiratory pressure of 5 cmH20,
* No scheduled surgery in the next 48 hours,
* Maximal inspiratory pressure < -20cmH20
* Airway occlusion pressure at 0.1 sec >6mmHg with a support pressure of 7 cmH20 and 0 cmH20 of positive end-expiratory pressure.

Exclusion Criteria:

* Scheduled neurosurgical surgery (duration of mechanical ventilation <24 hours),
* Neuromuscular disease,
* Spinal cord injury,
* Tracheostomy,
* Inability to be evaluated,
* Severe multiple injuries evaluated by the Injury Severity Score,
* Direct extubation and self-extubation,
* Patients who died during their ICU stay
* Patients transferred to another hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-09; Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALBERTO BELENGUER MUNCHARAZ, MD, Principal Investigator — Hospital General Universitario de Castellón
Locations (1):
- Hospital General Universitario Castello, Castelló, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belenguer-Muncharaz A, Diaz-Tormo C, Granero-Gasamans E, Mateu-Campos ML. Protocol-directed weaning versus conventional weaning from mechanical ventilation for neurocritical patients in an intensive care unit: a nonrandomized quasi-experimental study. Crit Care Sci. 2023 Mar 1;35(1):44-56. doi: 10.5935/2965-2774.20230340-en. PMID 37712729

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Protocol-directed Weaning | Conventional Weaning
Started | 50 | 44
Completed | 50 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Protocol-directed Weaning | Conventional Weaning | Total
Number analyzed (Participants) | 50 | 44 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 31 | 23 | 54
  >=65 years | 17 | 20 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (19) | 58 (19) | 56 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 30 | 27 | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 50 | 44 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Extubation Failure
Description: Rate of failure after extubation (increase of respiratory rate, deterioration of oxygenation, increase of cardiac rate or blood pressure)
Time Frame: 2 days after extubation
Population: In conventional group, 9 participants were tracheostomized directly without previous extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Protocol-directed Weaning | Conventional Weaning
Number analyzed (Participants) | 50 | 35
Participants | 8 | 6

2. Secondary Outcome: Number of Participants With Need for Tracheostomy
Description: Need for tracheostomy during process of weaning either before or after extubation
Time Frame: Along intensive care unit stay (30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Protocol-directed Weaning | Conventional Weaning
Number analyzed (Participants) | 50 | 44
Participants | 4 | 11

3. Secondary Outcome: Duration of Mechanical Ventilation
Description: Measure all the time (in days) the patient is connected to mechanical ventilation
Time Frame: Intensive Care unit stay (30 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Protocol-directed Weaning | Conventional Weaning
Number analyzed (Participants) | 50 | 44
days | 5 [2 to 13] | 9 [3 to 22]

4. Secondary Outcome: Intensive Care Unit Stay
Description: Measure length of stay at intensive care unit
Time Frame: days (30 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Protocol-directed Weaning | Conventional Weaning
Number analyzed (Participants) | 50 | 44
days | 9 [5 to 20] | 14 [6 to 29]

5. Secondary Outcome: Hospital Stay
Description: Measure length of stay at hospital
Time Frame: days (2 months)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Protocol-directed Weaning | Conventional Weaning
Number analyzed (Participants) | 50 | 44
days | 24 [17 to 48] | 33 [19 to 52]

6. Secondary Outcome: Intensive Care Unit Mortality
Description: Mortality at intensive care unit
Time Frame: Along intensive care unit stay (30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Protocol-directed Weaning | Conventional Weaning
Number analyzed (Participants) | 50 | 44
Participants | 4 | 3

7. Secondary Outcome: Hospital Mortality
Description: Mortality at hospital (including at intensive care unit)
Time Frame: Along hospital stay (2 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Protocol-directed Weaning | Conventional Weaning
Number analyzed (Participants) | 50 | 44
Participants | 5 | 8

8. Secondary Outcome: 90-day Mortality
Description: Mortality at 90 days after inclusion at study
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Protocol-directed Weaning | Conventional Weaning
Number analyzed (Participants) | 50 | 44
Participants | 6 | 9

ADVERSE EVENTS:
Time Frame: - Serious adverse events were not monitored/assessed during study period (until 90 days after inclusion). - Not serious adverse events were not monitorized/assessed during study period (until 90 days after inclusion). - All-cause mortility was monitorized/assessed in outcomes measurements: ICU mortality, hospital mortality and 90-day mortality
Description: * Serious, and other [Not Including Serious] adverse events were not monitored/assessed.
  * All-cause mortality has been registered in outcome measurements: ICU Mortality, Hospital Mortality and 90-d Mortality.
Arm/Group | Protocol-directed Weaning | Conventional Weaning
All-Cause Mortality (participants affected / at risk) | 6/50 | 9/44
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT03128086/Prot_SAP_000.pdf